CLINICAL TRIAL: NCT05275478
Title: A Phase 1/2, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, and Preliminary Anti-tumor Activity of TNG908 in Patients With MTAP-deleted Advanced or Metastatic Solid Tumors
Brief Title: Safety and Tolerability of TNG908 in Patients With MTAP-deleted Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tango Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TNG908-C101
Record Dates: First submitted 2022-02-18; First posted 2022-03-11 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Solid Tumor
Keywords: MTAP deletion; PRMT5; cholangiocarcinoma; NSCLC; mesothelioma; MPNST; Tango; Glioblastoma multiforme; pancreatic; GBM; sarcoma
MeSH Terms: conditions — Cholangiocarcinoma; Mesothelioma; Neurofibrosarcoma; Glioblastoma; Sarcoma

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation (sequential) followed by phase 2 dose expansion in 6 arms (parallel)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Escalation (Experimental): Participants with MTAP-deleted solid tumors will receive escalating doses of TNG908 to estimate the MTD
  Interventions: Drug: TNG908
- Dose Expansion in NSCLC (Experimental): Participants with MTAP-deleted NSCLC (squamous and non squamous) will receive TNG908 at the identified RP2D
  Interventions: Drug: TNG908
- Dose Expansion in Mesothelioma (Experimental): Participants with MTAP-deleted mesothelioma will receive TNG908 at the identified RP2D
  Interventions: Drug: TNG908
- Dose Expansion in Pancreatic Ductal Adenocarcinoma (Experimental): Participants with MTAP-deleted pancreatic ductal adenocarcinoma will receive TNG908 at the identified RP2D
  Interventions: Drug: TNG908
- Dose Expansion in Sarcoma (Experimental): Participants with MTAP-deleted sarcoma (soft tissue and bone) will receive TNG908 at the identified RP2D
  Interventions: Drug: TNG908
- Dose Expansion in solid tumors (Experimental): Participants with other MTAP-deleted solid tumors will receive TNG908 at the identified RP2D
  Interventions: Drug: TNG908
- Dose Expansion in Glioblastoma (Experimental): Participants with MTAP-deleted relapsed/refractory glioblastoma will receive TNG908 at the identified RP2D
  Interventions: Drug: TNG908

INTERVENTIONS:
Drug: TNG908 — TNG908, a selective PRMT5 inhibitor, will be administered orally

SUMMARY:
This is a first in human study in patients with advanced or metastatic solid tumors known to have an MTAP deletion. The first part of the study is an open-label, dose escalation and the second part is an open label dose expansion in specific MTAP-deleted tumor types. The study drug, TNG908, is a selective PRMT5 inhibitor administered orally. The study is planned to treat up to 192 participants.

DETAILED DESCRIPTION:
This is a Phase 1/2 multi-center, open label study in solid tumor patients (including glioblastoma) who have a confirmed homozygous MTAP deletion in their tumor. The Phase 1 portion is a dose escalation study of oral TNG908 in patients with confirmed MTAP-deleted solid tumors. In Phase 2, 6 expansion arms defined by confirmed MTAP-deleted tumor types will enroll in parallel at the RP2D of TNG908. In both parts of the study participants who tolerate the drug may continue treatment until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years-of-age at the time of signature of the main study ICF
2. Performance status: ECOG Performance Score of 0 to 1 or Karnofsky performance status score ≥70.
3. Confirmed histologic or cytologic diagnosis of a locally advanced, metastatic, and/or unresectable solid tumor or for GBM, have R/R disease.
4. Prior standard therapy, as available
5. Documented bi-allelic (homozygous) deletion of MTAP in a tumor detected by next- generation sequencing or absence of MTAP protein in a tumor detected by IHC.
6. Adequate organ function/reserve per local labs
7. Adequate liver function per local labs
8. Adequate renal function per local labs
9. Negative serum pregnancy test result at screening
10. Written informed consent must be obtained according to local guidelines

Exclusion Criteria:

1. Known allergies, hypersensitivity, or intolerance to TNG908 or its excipients
2. Uncontrolled intercurrent illness that will limit compliance with the study requirements
3. Active infection requiring systemic therapy
4. Currently participating in or has planned participation in a study of another investigational agent or device
5. Impairment of GI function or disease that may significantly alter the absorption of oral TNG908
6. Active prior or concurrent malignancy.
7. Central nervous system metastases associated with progressive neurological symptoms
8. Current active liver disease from any cause
9. Known to be HIV positive, unless all of the following criteria are met:

   1. CD4+ count ≥300/μL
   2. Undetectable viral load
   3. Receiving highly active antiretroviral therapy
10. Clinically relevant cardiovascular disease
11. A female patient who is pregnant or lactating
12. Patient is unwilling or unable to comply with the scheduled visits, drug administration plan, laboratory tests, biopsy, or other study procedures and study restrictions
13. Patient has a prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion, may affect the safety of the patient or impair the assessment of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: | 28 days
  To determine the MTD and dosing schedule of TNG908
Phase 2: | 16 weeks
  To assess anti-neoplastic activity of TNG908 in patients with MTAP-deleted advanced solid tumors by RECIST or mRECIST v1.1 or modified RANO criteria

SECONDARY OUTCOMES:
Phase 1: | 16 weeks
  To assess preliminary evidence of anti-neoplastic activity of TNG908 in patients with MTAP-deleted advanced solid tumors by RECIST or mRECIST v1.1or modified RANO criteria
Phase 1 and 2: | 28 days
  To describe the safety and tolerability profile of TNG908 by frequency and severity of AEs
Phase 1 and 2: | 16 days
  Area under the plasma concentration versus time curve (AUC)
Phase 1 and 2: | 16 days
  Time to achieve maximal plasma concentration (Tmax)
Phase 1 and 2: | 16 days
  Maximum observed plasma concentration (Cmax)
Phase 1 and 2: | 16 days
  Terminal elimination half-life (t1/2)
Phase 1 and 2: | 16 days
  Apparent total plasma clearance when dosed orally (CL/F)
Phase 1 and 2: | 16 days
  Apparent volume of distribution when dosed orally (Vz/F)
Phase 1 and 2: | 28 days
  SDMA levels in tumor tissue will be assessed pre-treatment and post treatment with TNG908

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Pimkin, MD, PhD, Study Director — Tango Therapeutics, Inc.
Locations (20):
- United States (15):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Florida Cancer Specialists & Research Institute, Lake Mary, Florida
  - Northwestern University, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, Fairfax, Virginia
- France (5):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - EDOG Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Institut Oncopole Claudius Regaud, Toulouse
  - Institute Gustav Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Briggs KJ, Cottrell KM, Tonini MR, Tsai A, Zhang M, Whittington DA, Zhang W, Lombardo SA, Yoda S, Wilker EW, Meier SR, Yu Y, Teng T, Huang A, Maxwell JP. TNG908 is a brain-penetrant, MTA-cooperative PRMT5 inhibitor developed for the treatment of MTAP-deleted cancers. Transl Oncol. 2025 Feb;52:102264. doi: 10.1016/j.tranon.2024.102264. Epub 2025 Jan 4. PMID 39756156